CLINICAL TRIAL: NCT02162706
Title: Pilot Study of Salivary Cortisol Measurements by Mass Spectrometry
Brief Title: Salivary Cortisol Measurements by Mass Spectrometry
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tandy Aye, Associate Professor, Stanford University
Other Study IDs: Salivary Cortisol
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Endocrine Disorders
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Saliva was collected using Salivabio children's swab (SCS).
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Non intervention study

SUMMARY:
Cortisol is a hormone critical for survival in times of stress. Currently most measurements are done with blood samples. The hypothesis of this study is cortisol measured from saliva using mass spectrometry can be used to replace measurements by blood.

DETAILED DESCRIPTION:
Cortisol levels change depending on the time of day. Salivary samples were collected from health controls at bedtime, midnight and first morning waking on two consecutive nights and salivary cortisol levels were measured using mass spectrometry. In a patients with possible endocrine disorders who were going through an adrenocortiotropin stimulation test for adrenal insufficiency, salivary cortisol was measured prior to giving cosyntropin and 30-40 minutes after cosyntropin.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects
* Subjects with possible endocrine disorder

Exclusion Criteria:

* Tracheostomy or ventilator dependent
* Gastrotomy tubed dependent or unable to eat/drink by mouth

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with possible endocrine disorders seen during outpatient pediatric endocrinology visit or inpatient consultations. Healthy controls were open to the general public in California.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol | All collections are done within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tandy Aye, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital and Stanford Clinics, Stanford, California, United States

REFERENCES:
- [Background] Deutschbein T, Unger N, Mann K, Petersenn S. Diagnosis of secondary adrenal insufficiency: unstimulated early morning cortisol in saliva and serum in comparison with the insulin tolerance test. Horm Metab Res. 2009 Nov;41(11):834-9. doi: 10.1055/s-0029-1225630. Epub 2009 Jul 7. PMID 19585406
- [Background] Baid SK, Sinaii N, Wade M, Rubino D, Nieman LK. Radioimmunoassay and tandem mass spectrometry measurement of bedtime salivary cortisol levels: a comparison of assays to establish hypercortisolism. J Clin Endocrinol Metab. 2007 Aug;92(8):3102-7. doi: 10.1210/jc.2006-2861. Epub 2007 Jun 5. PMID 17550962
- [Result] Chao CS, Shi RZ, Kumar RB, Aye T. Salivary cortisol levels by tandem mass spectrometry during high dose ACTH stimulation test for adrenal insufficiency in children. Endocrine. 2020 Jan;67(1):190-197. doi: 10.1007/s12020-019-02084-8. Epub 2019 Sep 18. PMID 31535345